CLINICAL TRIAL: NCT00860990
Title: VA GI Quality of Life Survey
Brief Title: VA Gastrointestinal (GI) Quality of Life Survey
Acronym: VA GI QOL
Status: Terminated | Type: Observational
Why Stopped: Outcome measures are included in another, similar study.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Korsten, Mark - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: B4162C-4; 2380-07-042
Record Dates: First submitted 2009-03-06; First posted 2009-03-13 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: SCI

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: SCI or disabled
  Interventions: Other: Completion of GI quality of life survey
- 2: Able-bodied
  Interventions: Other: Completion of GI quality of life survey

INTERVENTIONS:
Other: Completion of GI quality of life survey — Subjects are asked to complete a survey related to bowel care and its effects on various variables related to quality of life.

SUMMARY:
Spinal cord injury (SCI) often results in reduced bowel function and regularity, leading to a decrease in quality of life for those who are affected. Evidence-based research has indicated that, when surveyed, individuals with SCI express a greater reduction in quality of life derived from their bowel routine than able-bodied subjects. In addition, the extent of reduction in quality of life has a direct relationship with the level of Injury. Those with tetraplegia score worse than those with paraplegia and paraplegics score worse than controls. The development of an adequate quality of life questionnaire is needed to effectively identify the impact of bowel care on quality of life in patients with SCI compared to able-bodied controls. The purpose of this study is to determine the discriminatory ability of the survey for various diagnoses such as SCI, CVA, TBI, chronic back pain, radiculopathy from the Rehabilitation Service and able bodied persons.

DETAILED DESCRIPTION:
In an abstract " A Bowel Care Survey to Assess Quality of Life in Persons With Spinal Cord Injury" in Journal of Spinal Cord Medicine in 2006, JP Lirio, et al surveyed 20 subjects (10 controls, 5 para, 5 tetra). The survey consisted of 42 items relating to GI function, bowel program/routine and quality of life. Survey items were weighted across a range of outcomes (e.g., complete continence=0 to frequent incontinence of solid evacuate=5). Total survey scores were compared among the groups by ANOVA with a Scheffe post hoc test. In those with SCI, level of injury (LOI) was converted to a numeric value and the relationship between LOI and total score was determined by simple regression.

The range of scores across the groups was 2 to 111 points. The controls scored significantly lower than those in the Para group who were significantly lower than those in the Tetra group (6 5 vs. 46 38 vs. 92 24, P<0.01, respectively). Within SCI, 43% of the variance of the total score was explained by level of injury. (r2=42.5, P<0.05), which is suggestive for the potential of good content validity of this tool. The authors concluded that the preliminary results of this survey show that persons with greater degrees of neurological impairment also manifest a greater negative impact from bowel care on their QoL. These results are encouraging for being able to develop a sensitive tool that will capture changes in bowel care status after therapeutic intervention that would be expected to influence QoL.

Innovative and potentially efficacious treatments for bowel care are being developed. There is a clinical/investigative need for a valid survey that is sensitive to quality of life (QoL) changes relating to interventions for bowel care in those with spinal cord injury (SCI). This is an ongoing project to develop a self-reported gastrointestinal (GI) survey that measures the impact of bowel function on QoL in individuals with SCI. This research seeks to develop a quality of life questionnaire that can be used to assess bowel function in able bodied individuals as well as spinal cord patients. This tool is essential for measuring change in bowel function due to an intervention or aging, rehabilitation, medications, etc.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Able to understand English

Exclusion Criteria:

* Diagnosed dementia, severe TBI or other conditions which limit the ability to provide acute information in the judgment of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers will be recruited from the spinal cord injury service/clinic, the primary care service/clinic, the geriatric service/clinic, the chronic kidney service/clinic, and the rehabilitation service/clinic at the James J. Peters VA Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Quality of life relative to bowel function and care | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Korsten, MD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States